CLINICAL TRIAL: NCT06453226
Title: PArkinson's Non-Invasive Volatile ORganic Compound Analysis and Microbiome Assessment (PANORAMA) Study
Brief Title: Non-invasive Detection of Volatile Metabolites in Parkinson's Disease
Acronym: PANORAMA
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 311577; 22/NI/0090 (Other: REC)
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: volatile organic compounds
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's group: Patients with confirmed Parkinson's disease undergoing neurological examination
- Healthy Controls: Patients will be asked to nominate a partner/carer that can be enrolled in the control group. Healthy controls will also be recruited using web-based adverts mainly via the Imperial Clinical Research Facility and Parkinson's disease charities.
- De-Novo: Patients undergoing neurological examination for suspected Parkinson's disease due to presence of symptoms

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder. Currently, a diagnostic test for early PD does not exist.

The aim to address this problem by developing a non-invasive breath test to differentiate early PD from controls. Small molecules contained in breath, which offers precious information about disease presence, will be analysed. Data from the breath molecules and gut bacterial changes occurring in PD will be combined. These bacterial changes have been shown to arise years before the development of PD symptoms.

Thanks to earlier diagnosis, therapies could start in advance and improve clinical outcomes and quality of life.

DETAILED DESCRIPTION:
Detection of volatile organic compounds (VOCs) within exhaled breath and other biological matrices (such as urine, blood, saliva and skin) offers an attractive new strategy for non-invasive screening, diagnosis and monitoring of diseases. VOCs emitted by the body potentially reflect biochemical processes underlying physio-pathological states (Smith 2007). Non-invasive breath tests are well-accepted by patients, and for this reason they can offer the opportunity of large population screening and early diagnosis that can be crucial for several diseases (Belluomo 2021; Woodfield 2021). Despite breath testing has been proved effective to identify different disease states, among which cancer (Woodfield 2022) and infections (Kamal 2021), its application to neurodegenerative diseases remains still poorly explored.

Parkinson's disease (PD) is one of the most common neurodegenerative disorders, with six million people affected worldwide and an incidence rate in rapid increase (Armstrong 2020). Currently, diagnosis of PD is based primarily on the presence of specific motor symptoms, such as bradykinesia, rigidity and rest tremor, which manifest when the progressive accumulation of Lewy body pathology and loss of melanised dopaminergic neurons in the substantia nigra pars compacta is already in a mid-late stage (Armstrong 2020). Misdiagnosis is common on clinical criteria alone, particularly at early presentation when symptoms overlap with other Parkinson-Plus syndromes and secondary Parkinsonism conditions (Rizzo 2016). Identification of novel biomarkers could lead to earlier and more accurate diagnoses and consequently remarkably improve patient management and quality of life.

It is hypothesised that specific VOC signatures differentiate PD patients from healthy controls. The microbiome alterations found in PD could be at the origin of VOC decreased or increased production.

The study recruitment will comprise patients with PD (50), healthy controls (mainly patient's partners or carers 50), and 20 de-novo not medicated PD patients. Different tyoes of samples will be collected (i) breath for volatile organic compound analysis (ii) stool for microbiome characterisation and (iii) blood for microvesicles extraction.

ELIGIBILITY:
Inclusion Criteria [PD group]:

* (i) Patients undergoing neurological examination for confirmed or suspected Parkinson's disease
* (ii) Patients aged ≥18 years and below 90 years of age;
* (iii) Patients off antibiotic or probiotic therapies for at least the last 4 weeks;
* (iv) Patients without formal diagnosis of dysbiotic conditions;
* (v) Patients with capacity.

Inclusion Criteria [Healthy Volunteers]:

* (i) healthy volunteers that may be or not partner or carer of a Parkinson's patient;
* (ii) Subject aged ≥18 years and below 90 years of age;
* (iii) Patients off antibiotic or probiotic therapies for at least the last 4 weeks;
* (iv) Patients without formal diagnosis of dysbiotic conditions;
* (iiv) Subject with capacity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population for this study will be divided in three groups: (i) Parkinson patients (ii) healthy controls (iii) de-novo patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarker and measurement of their levels for the development of a non-invasive breath test for Parkinson's diagnosis | June 2025
  The primary outcome is the identification of biomarkers and measurement of their levels in breath for the future development of a non-invasive breath test, able to diagnose Parkinson's disease. These levels will be measured using gas chromatography mass spectrometry. Differences will be identified in Parkinson's group vs de-novo and healthy controls and important compounds will be therefore identified.

SECONDARY OUTCOMES:
Characterisation of microbiome in Parkinson patients, de novo and healthy controls | June 2025
  Microbiome will be characterised in stool samples from the three study groups to identify differences due to Parkinson's. The bacteria type will be then linked to the VOC found in breath, to define if the VOC found in breath to differentiate Parkinson's patients from de novo and controls have a microbial origin.

CONTACTS AND LOCATIONS:
Locations (1):
- Charing Cross Hospital, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided